CLINICAL TRIAL: NCT06132802
Title: Evaluation of Anterior Repositioning Guided Splint Combined With or Without Injectable Platelet-rich Fibrin in Treatment of TMJ Internal Derangement.
Brief Title: Evaluation of Anterior Repositioning Guided Splint Combined With or Without I Platelet-rich Fibrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Mohammed Mahmoud Nasef (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Mohammed Mahmoud Nasef, Demonstrator at the Department of oral and Maxillofacial Surgery, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUAREC20210100-07
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Anterior repositioning guided splint; Injectable platelet-rich fibrin
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Arthrocentesis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: Patients who received treatment involving ARS and arthrocentesis only (Experimental)
  Interventions: Procedure: Patients who received treatment involving ARS and arthrocentesis only
- Group II: Patients who received treatment involving ARS, arthrocentesis, and an I-PRF injection (Experimental)
  Interventions: Procedure: Patients who received treatment involving ARS, arthrocentesis, and an I-PRF injection

INTERVENTIONS:
Procedure: Patients who received treatment involving ARS and arthrocentesis only — A 5mm acrylic anterior repositioning splint (ARS) with maxillary coverage was crafted from alginate impressions. After arthrocentesis, the ARS was worn incrementally over six months, starting at two hours and reaching 14 hours daily. In the second week, wear time was continuous, increasing to 24 hours daily (excluding meals) until the sixth month. The ramp was removed in the seventh week. Follow-ups involved grinding the splint by 1mm every four weeks. Arthrocentesis included anesthesia, betadine prep, and using two 18-gauge needles to inject Ringer's lactate solution (100-200 cc) for joint lavage, freeing the disc by moving the lower jaw in various orientations.
  Arms: Group I: Patients who received treatment involving ARS and arthrocentesis only
Procedure: Patients who received treatment involving ARS, arthrocentesis, and an I-PRF injection — A 5mm acrylic anterior repositioning splint (ARS) was crafted from alginate impressions, secured with Adam's clasps on upper first molars. After arthrocentesis, patients wore the splint incrementally over six months, starting at two hours and reaching 24 hours daily (excluding meals). The ramp was removed in the seventh week, and follow-ups included grinding the splint by 1mm every four weeks until it reached 3mm, guided by articulating paper.
  Arthrocentesis involved administering anesthesia, prepping the area with betadine, and using two 18-gauge needles to inject 2-3 ml of Ringer's lactate solution for joint lavage. The lower jaw was moved to free the disc and release fibrous tissue. I-PRF preparation included centrifuging collected blood for 3 minutes at 700 rpm, and the resulting I-PRF was injected into the superior joint space of the lavaged joints.
  Arms: Group II: Patients who received treatment involving ARS, arthrocentesis, and an I-PRF injection

SUMMARY:
The study aims to evaluate clinically and radiographically the effectiveness of arthrocentesis and injection of I-PRF with wearing ARS in comparison to arthrocentesis and ARS only.

DETAILED DESCRIPTION:
The patient will be seated at a 45° angle with the head turned toward the unaffected side. After preparing and disinfecting the target site with betadine, two points will be marked over the affected joint. Local anesthesia will be administered to block the auriculotemporal nerve. Using 19-gauge needles, the superior joint space will be distended with 2-3 ml of Ringer's solution. Another needle will be inserted into the distended compartment near the articular eminence to facilitate solution flow. Lactated Ringer's solution, connected to one needle, will be infused with sufficient pressure (200 mL in 15-20 minutes) to release adhesions. Following the removal of one needle, 2 ml of injectable platelet-rich fibrin (PRF) will be injected into the superior joint space.

For the preparation of injectable PRF, 20 ml of the patient's blood will be drawn and divided into two 10 ml vaccutainers. After centrifugation, the obtained PRF will be aspirated into a 5 ml syringe, and 1.5 to 2 ml of PRF will be injected into the superior joint space.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* History of unilateral or bilateral disc displacement without reduction (DDwoR) of the temporomandibular joint (TMJ) confirmed by MRI.
* Presence of TMJ pain and restricted maximum mouth opening.
* No improvement with conservative treatment.
* Absence of MRI contraindications.

Exclusion Criteria:

* Patients having any systemic disease that could interfere with the TMJ treatment or assessment.
* Patients having previous TMD treatment modalities or previous TMJ surgery.
* Patients with a previous history of oral and or maxillofacial trauma.
* Patients that are contraindicated to perform MRI.
* Completely or partially edentulous patients were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Maximum mouth opening | First week, first month, third months, and sixth months
  Maximum Mouth Opening was determined by measuring the distance between the incisal edges of the upper and lower incisors. In Millimeter (mm)
Pain score | First week, first month, third months, and sixth months
  Using Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Right and left lateral excursion | First week, first month, third months, and sixth months
  In Millimeter (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine Al-Azhar University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Yuce E, Komerik N. Comparison of the Efficiacy of Intra-Articular Injection of Liquid Platelet-Rich Fibrin and Hyaluronic Acid After in Conjunction With Arthrocentesis for the Treatment of Internal Temporomandibular Joint Derangements. J Craniofac Surg. 2020 Oct;31(7):1870-1874. doi: 10.1097/SCS.0000000000006545. PMID 32433129
- [Background] Herrera-Vizcaino C, Dohle E, Al-Maawi S, Booms P, Sader R, Kirkpatrick CJ, Choukroun J, Ghanaati S. Platelet-rich fibrin secretome induces three dimensional angiogenic activation in vitro. Eur Cell Mater. 2019 Apr 9;37:250-264. doi: 10.22203/eCM.v037a15. PMID 30963526
- [Background] Teama UA. Evaluation of Injectable platelet rich fibrin for the management of Tempromandibular joint internal derangement.(clinical evaluation). Egy Dent J. 2020; 66:883-91.
- [Background] Marzook HAM, Abdel Razek AA, Yousef EA, Attia AAMM. Intra-articular injection of a mixture of hyaluronic acid and corticosteroid versus arthrocentesis in TMJ internal derangement. J Stomatol Oral Maxillofac Surg. 2020 Feb;121(1):30-34. doi: 10.1016/j.jormas.2019.05.003. Epub 2019 May 20. PMID 31121331
- [Background] AbdulRazzak NJ, Sadiq JA, Jiboon AT. Arthrocentesis versus glucocorticosteroid injection for internal derangement of temporomandibular joint. Oral Maxillofac Surg. 2021 Jun;25(2):191-197. doi: 10.1007/s10006-020-00901-3. Epub 2020 Sep 1. PMID 32870434